CLINICAL TRIAL: NCT02851784
Title: Combination Therapy of Microwave Ablation and Expanding Activated Autologous Lymphocytes for Hepatocellular Carcinoma
Brief Title: Combination Therapy of Microwave Ablation and Cellular Immunotherapy for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: liangping
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; ablation; immunotherapy; cytokine induced kill cell
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MWA only (Active Comparator): The HCC patients will be treated only by MWA.No adoptive immunotherapy will be used.
  Interventions: Procedure: MWA
- MWA combined with immunotherapy (Experimental): The HCC patients will be treated firstly by MWA, and then treated by courses of adoptive immunotherapy.
  Interventions: Biological: adoptive immunotherapy; Procedure: MWA

INTERVENTIONS:
Biological: adoptive immunotherapy — HCC (D ≤5 cm, fewer than three tumors) patients were treated with radical MWA and 4-6 courses of immunotherapy with CIK every year.The immunotherapy were started at 2 weeks, 4 weeks, 6 weeks, 10 weeks, 14 weeks, 18 weeks and then every 12 weeks after MWA. Peripheral blood mononuclear cells were differentiated into phenotypically confirmed DCs and effector cells. DC-CIK and CTL were injected into the abdominal cavity. CIK was infused intravenously.
  Other Names: cytokine induced kill cell
  Arms: MWA combined with immunotherapy
Procedure: MWA — ALL the HCC patients will be treated only by microwave ablation and then enter the follow-up

SUMMARY:
The study is to observe safety, survival effect and peripheral T-lymphocyte subsets of combination therapy with percutaneous microwave ablation (MWA) and adoptive immunotherapy in hepatocellular carcinoma(HCC).

DETAILED DESCRIPTION:
HCC (D ≤5 cm, fewer than three tumors) patients were treated with radical MWA and 4-6 courses of immunotherapy with CIK every year. The immunotherapy were started at 2 weeks, 4 weeks, 6 weeks, 10 weeks, 14 weeks, 18 weeks and then every 12 weeks after MWA. Peripheral blood mononuclear cells were differentiated into phenotypically confirmed DCs and effector cells. DC-CIK and CTL were injected into the abdominal cavity. CIK was infused intravenously. The safety, survival effect and peripheral T-lymphocyte subsets of combination therapy group will be recorded and compared with those of MWA group.

ELIGIBILITY:
Inclusion Criteria:

1. single HCC of 5 cm or smaller;
2. three or fewer multiple HCC with a maximum dimension of 3 cm or less;
3. absence of portal vein thrombosis or extrahepatic metastases;
4. Child-Pugh classification A or B;
5. tumor accessible via a percutaneous approach. white blood cell count >2 x 109/L, platelet count >40 x 109/L,serum creatinine <110 μmol/L, aspartate aminotransferase <3 times the upper limit, serum bilirubin <2.5 times the upper limit, prothrombin time <19 seconds.

Exclusion Criteria:

1. pregnant or breast-feeding; psychiatric problems, addiction, or any other disorder that prevented informed consent;
2. active uncontrolled infection; concurrent systemic corticosteroid treatment;
3. systemic autoimmune disease;
4. clinically significant ischemic heart disease or cardiac failure;
5. and chemotherapy or radiotherapy within the preceding 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Cumulative survival rates were calculated by the Kaplan-Meier method, and comparison between MWA and combination treatment will be done by the log-rank test. | up to 8 years

SECONDARY OUTCOMES:
disease free survival rates were calculated by the Kaplan-Meier method, and comparison between MWA and combination treatment will be done by the log-rank test | up to 8 years

OTHER OUTCOMES:
Local tumor progress rates were calculated by the Kaplan-Meier method, and comparison between MWA and combination treatment will be done by the log-rank test | up to 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Dr., Study Director — Chinese PLA General Hospial
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided